CLINICAL TRIAL: NCT03130335
Title: Intra-articular Autologous Bone Marrow Aspirate Injection for the Treatment of Knee Osteoarthritis: a Pilot Study With Radiological Follow-up
Brief Title: Intra-articular Autologous Bone Marrow Aspirate Injection for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0435
Record Dates: First submitted 2017-04-20; First posted 2017-04-26 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — cyclomaltodextrin glucanotransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Marrow Aspirate (BMA) Injection (Experimental)
  Interventions: Procedure: BMA Injection; Biological: BMA

INTERVENTIONS:
Procedure: BMA Injection — Bone marrow will be aspirated from the iliac crest and injected into the knee.
Biological: BMA — Bone marrow will be aspirated from the iliac crest.

SUMMARY:
Knee osteoarthritis (OA) is a leading cause of disability. The objectives of treatment are to reduce pain, improve function, and slow down further breakdown of the knee. Recently, research on nonsurgical treatment options for knee OA has increased significantly. One potential treatment of interest is the use of stem cell injections. Stem cells are one's own cells that have the ability to divide into other types of cells, and may cause regrowth of cartilage when injected into the knee. There have been few, but promising, studies that show improvements in pain and function with stem cell injections in those with knee OA. Therefore, more research is needed to identify patients who might benefit from this injection. This pilot study will look at changes in pain and function for 20 patients at 1, 3, 6, and 12 months after a stem cell injection into the knee. Patients will also undergo magnetic resonance imaging at 6 months and 12 months following the injection.

ELIGIBILITY:
Inclusion Criteria:

* >=3 months of symptomatic knee OA unresponsive to at least two of the following: activity modification, physical therapy, bracing, assistive devices, acupuncture, non-steroidal anti-inflammatory medications, local steroid injections, and hyaluronic acid injections
* Radiographically confirmed Kellgren-Lawrence I-II knee OA (mild knee OA; no bone-on-bone)
* Age 18-79 years

Exclusion Criteria:

* Presence of loose bodies on baseline magnetic resonance imaging
* Clinically and radiologically confirmed anterior/posterior cruciate ligament deficiences
* History of meniscal injury other than degenerative meniscal tears
* Previous knee surgery
* Presence of a degenerative meniscal tear causing mechanical symptoms such as locking, buckling, or give-way
* Intra-articular injection to affected knee within 6 weeks of intra-articular BMA injection
* Mechanical axis deviation greater than 7 degrees
* Intolerance to acetaminophen or hydrocodone (i.e., Vicodin)
* Use of non-steroidal anti-inflammatory drugs <1 weeks prior to BMA
* Injection of the joint scheduled for treatment within 3 months of BMA injection
* Body mass index of 30 or more
* History of drug abuse
* Current cigarette smokers
* Current use of systemic steroids
* History of or current alcohol abuse or dependence
* History of anemia, bleeding disorders, or inflammatory joint disease
* Active infection
* Active malignancy per medical or surgical history, diagnosed by primary case physician or treating specialist, undergoing treatment, has undergone treatment, or has declined treatment
* Inability to refrain from statin regimen from 1 month pre-injection to 1 month post-injection
* Pregnancy or breastfeeding at time of treatment
* Participating or planning to participate in a worker's compensation program at the time of treatment or follow-up period
* Pending or planned legal action pertaining to knee pain
* Non-English speaking

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Jr. | 1 month after date of injection
  The KOOS Jr. measures patient-reported pain and function. The score ranges from 0-100, with 0 representing total knee disability and 100 representing perfect knee health.
KOOS Jr. | 3 months after date of injection
  The KOOS Jr. measures patient-reported pain and function. The score ranges from 0-100, with 0 representing total knee disability and 100 representing perfect knee health.
KOOS Jr. | 6 months after date of injection
  The KOOS Jr. measures patient-reported pain and function. The score ranges from 0-100, with 0 representing total knee disability and 100 representing perfect knee health.
KOOS Jr. | 12 months after date of injection
  The KOOS Jr. measures patient-reported pain and function. The score ranges from 0-100, with 0 representing total knee disability and 100 representing perfect knee health.

SECONDARY OUTCOMES:
Pain | 1 month, 3 months, 6 months, and 12 months after date of injection
  Pain will be assessed using the numerical rating scale (NRS), which is on a scale of 0-10. 10 represents worst pain, and 0 represents no pain.
Degree of cartilage change | 6 months (first 5 patients only) and 12 months after date of injection
  Cartilage change will be assessed via magnetic resonance imaging.
Presence of side effects | 1 month, 3 months, 6 months, and 12 months after date of injection
  The presence of side effects, including increased pain, bleeding, infection, and motor-sensory deficits, will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Lutz, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Wells K, Klein M, Hurwitz N, Santiago K, Cheng J, Abutalib Z, Beatty N, Lutz G. Cellular and Clinical Analyses of Autologous Bone Marrow Aspirate Injectate for Knee Osteoarthritis: A Pilot Study. PM R. 2021 Apr;13(4):387-396. doi: 10.1002/pmrj.12429. Epub 2020 Jul 13. PMID 32500620